CLINICAL TRIAL: NCT05920278
Title: Performance of the Movano Health Ring in a Controlled Hypoxia Study: Prospective Observational Study
Brief Title: Accuracy of Pulse Oximeters in Profound Hypoxia
Status: Completed | Type: Observational
Sponsor: Movano Health (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 153-00381
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2023-06

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Adult Volunteers: Minimum of ten (10) subjects meeting the eligibility criteria.
  Interventions: Device: Pulse oximeter

INTERVENTIONS:
Device: Pulse oximeter — Devices (2) were placed on the finger and the fingertip. Blood samples were taken at each stable level of oxygenation.

SUMMARY:
The goal of this study was to evaluate the accuracy of pulse oximeters over the range of 70-100%. Two devices were placed on each subject with one on the finger and the other on the fingertip. SpO2 measurements from these devices were compared to sampling of arterial blood during brief stable oxygen desaturation in healthy volunteers to evaluate the claimed range.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good general health with no evidence of any medical problems.
* Subject is fluent in both written and spoken English.
* Subject provided written informed consent and is willing to comply with the study procedures.
* Subject is willing to have their skin color assessed.

Exclusion Criteria:

* Subject is obese with a BMI over 30.
* Subject has a known history of heart disease, lung disease, kidney or liver disease.
* Subject has asthma, sleep apnea, or uses a CPAP.
* Subject has diabetes.
* Subject has a clotting disorder, anemia, or in the opinion of the investigator, they would be unsuitable for participation.
* Subject has any other serious system illness.
* Subject is a current smoker.
* Subject has any injury, deformity, or abnormality at the sensor sites that, in the opinion of the investigator, would interfere with the sensors working correctly.
* Subject has a history of fainting or vasovagal response.
* Subject has a sensitivity to local anesthesia.
* Subject has Raynaud's disease.
* Subject has unacceptable collateral circulation based on an exam by the investigator.
* Subject is pregnant, lactating, or trying to get pregnant.
* Subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with the study procedures.
* Subject has any other condition, which in the opinion of the investigator, would make them unsuitable for the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult participants 18 to 49 years old, of which 2 or 15% of the subject pool is darkly pigmented.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
RMSE compared to arterial blood SaO2 | 2 days
  Root Mean Squared Error between Movano Ring SpO2 measurement and the arterial blood SaO2 calibrated using arterial blood gas.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip E Bickler, MD, PhD, Principal Investigator — University of California at San Francisco (UCSF)
Locations (1):
- Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mastrototaro JJ, Leabman M, Shumate J, Tompkins KL. Performance of a Wearable Ring in Controlled Hypoxia: A Prospective Observational Study. JMIR Form Res. 2024 Jun 5;8:e54256. doi: 10.2196/54256. PMID 38838332
- See also: Pulse Oximeters - Premarket Notification Submissions [510(k)s]: Guidance for Industry and Food and Drug Administration Staff | FDA — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/pulse-oximeters-premarket-notification-submissions-510ks-guidance-industry-and-food-and-drug